CLINICAL TRIAL: NCT06987773
Title: A Pivotal, Phase 1, Randomized, Open-Label, Single-Dose, Two-Way Crossover, Bioequivalence Study of Sapropterin Dihydrochloride 100 mg/mL Oral Suspension (Product Code: RLF-OD032) and Kuvan® (Sapropterin Dihydrochloride) 100 mg Powder for Oral Solution in Healthy Participants Under Fed Conditions
Brief Title: Study on Sapropterin Dihydrochloride Oral Suspension in Healthy Subjects Under Fed Conditions
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-5705
Record Dates: First submitted 2025-05-07; First posted 2025-05-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Suspensions; sapropterin; Powders; Solutions

STUDY DESIGN:
Intervention Model Description: Adaptative design
  In each period, subjects will receive one of the following treatments, according to the randomization scheme:
  Treatment A: 1 x 10 mg/kg dose of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  Treatment B: 1 x 10 mg/kg dose of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AB (Other): A) A single 10 mg/kg dose of a 100 mg/mL oral suspension of sapropterin dihydrochloride (RLF-OD032) , administered under fed conditions without water followed by B) A single 10 mg/kg dose of a 100 mg powder for oral solution of the Reference Product (Kuvan) , dissolved in water, administered under fed conditions with water
  Interventions: Drug: RLF-OD032 100 mg/mL oral suspension; Drug: Kuvan 100 MG Powder for Oral Solution
- BA (Other): B) A single 10 mg/kg dose of a 100 mg powder for oral solution of the Reference Product (Kuvan) , dissolved in water, administered under fed conditions with water followed by A) A single 10 mg/kg dose of a 100 mg/mL oral suspension of sapropterin dihydrochloride (RLF-OD032), administered under fed conditions without water
  Interventions: Drug: RLF-OD032 100 mg/mL oral suspension; Drug: Kuvan 100 MG Powder for Oral Solution

INTERVENTIONS:
Drug: RLF-OD032 100 mg/mL oral suspension — Sapropterin dihydrochloride
Drug: Kuvan 100 MG Powder for Oral Solution — Sapropterin dihydrochloride

SUMMARY:
This is a single center, Phase 1, randomized, open-label, single-dose, 2 treatment, 2-period,2-sequence, crossover study designed to compare the pharmacokinetics (PK) of sapropterin between the Test and Reference products in healthy Participants.

DETAILED DESCRIPTION:
In each period, subjects will receive a single 10 mg/kg dose of sapropterin dihydrochloride on Day 1, under fed conditions, followed by 24 hours of PK sampling.

The study will include a screening visit from Day -30 to Day -1. In each period, eligible subjects will be admitted to the clinical site on Day -1 and will be confined until completion of the assessments on Day 2. There will be a washout period of at least 7 days between doses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants, light smokers (no more than 10 cigarettes daily) or non-smokers, from 18 to 50 years of age.
2. BMI ≥18.5 and ≤30 kg/m2 and weight ≥50.0 and ≤100.0 kg for males and ≥45.0 and ≤100.0 kg for females
3. Females may be of childbearing or non-childbearing potential:

   * Childbearing potential:
   * Physically capable of becoming pregnant
   * Non-childbearing potential:
   * Surgically sterile (i.e., both ovaries removed, uterus removed, or bilateral tubal ligation) at least three (3) months prior to first drug administration; and/or;
   * Postmenopausal (no menstrual period for at least 12 consecutive months without any other medical cause and a FSH value consistent with being postmenopausal).
4. Willing to use acceptable, effective methods of contraception.
5. Able to tolerate venipuncture.
6. Be informed of the nature of the study and give written consent prior to any study procedure.

Exclusion Criteria:

1. History of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the participant or impact the validity of the study results.
2. Clinically significant illness and/or surgery.
3. Known or suspected carcinoma.
4. History of hypersensitivity or idiosyncratic reaction to sapropterin dihydrochloride or any other drug substances with similar activity.
5. History of or predisposition to seizure which, in the opinion of the Investigator, would jeopardize the safety of the participant or impact the validity of the study results.
6. History of upper gastrointestinal (GI) mucosal inflammation, esophagitis, gastritis, pharyngitis, or oropharyngeal pain, which, in the opinion of the Investigator, would jeopardize the safety of the participant or impact the validity of the study results.
7. History of abuse of medicinal product or drugs within the last three (3) years.
8. History of alcohol addiction requiring treatment.
9. History or presence of alcoholism within the last three (3) years. (>40 g ethanol/day or >10 units per week [one (1) unit =150 mL of wine, or 360 mL of beer, or 45 mL of 45% alcohol])
10. History of recreational use of soft drugs (such as marijuana) within one (1) month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within three (3) months prior to screening.
11. Use of St. John's wort within 30 days prior to the first drug administration.
12. History of clinically significant lactose, galactose, or fructose intolerance.
13. Presence of hepatic or renal dysfunction.
14. Presence of mouth piercings (object or hole), presence of non-removable dentures and orthodontic appliances (e.g., braces, retainers), or any other alteration to the mouth that may be deemed by the Investigator to compromise drug delivery.

    Note: Dental fillings, crowns, bridges, and implants are permitted as they are not considered to compromise drug delivery.
15. History of malabsorption within the last year or presence of clinically significant gastrointestinal (GI) disease.
16. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
17. Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
18. Positive test result for urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, phencyclidine, and tricyclic antidepressants).
19. Difficulty fasting or consuming high-fat, high-calorie or standard meals.
20. Regularly smokes more than 10 cigarettes per day within 6 months prior to the first drug administration.
21. Participants who received an implanted or injected (depot injection) medication, including hormonal contraceptives, within three (3) months prior to the first drug administration.
22. Females who:

    * Have discontinued or changed the use of implanted, intrauterine, intravaginal, or injected hormonal contraceptives within six (6) months prior to the first drug administration;
    * Have discontinued or changed the use of oral or patch hormonal contraceptives within one (1) month prior to the first drug administration;
    * Are pregnant (serum β-hCG consistent with pregnancy); or
    * Are breast-feeding.
23. Donation or loss of whole blood (including clinical trials):

    * ≥50 mL and <500 mL within 30 days prior to the first drug administration; or
    * ≥500 mL within 56 days prior to the first drug administration.
24. Donation of plasma within seven (7) days prior to dosing.
25. Participation in a clinical trial that involved administration of a biological product within 90 days prior to the first drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize participant safety or the integrity of the study results.
26. Participation in a clinical trial that involved administration of an investigational medicinal product, marketed drug or device within 30 days prior to the first drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize participant safety or the integrity of the study results.
27. On a special diet within 30 days prior to the first drug administration (e.g., liquid, protein, raw food diet).
28. Have had a tattoo or body piercing within 30 days prior to the first drug administration.
29. Have clinically significant findings in vital signs measurements and systolic blood pressure (SBP) <90 mmHg or >150 mmHg and diastolic blood pressure (DBP) <50 or >90 mmHg, or PR <50 or >100 bpm). Vitals signs may be repeated up to two (2) times, to determine if the values are significantly abnormal.
30. Have clinically significant findings in a 12-lead ECG. ECG readings may be repeated up to two times, to determine if the values are significantly abnormal.
31. Have clinically significant abnormal laboratory values. Laboratory tests may be repeated up to two (2) times, to determine if the values are significantly abnormal.
32. Have significant diseases.
33. Use of any of the following drugs within 30 days prior to drug administration:

    * Breast cancer resistance protein (BCRP) substrates (e.g., rosuvastatin);
    * Drugs affecting nitric oxide-mediated vasorelaxation (e.g., PDE-5 inhibitors, sildenafil, vardenafil, or tadalafil);
    * Folate synthesis inhibitors (e.g. methotrexate, valproic acid, phenobarbital, or trimethoprim);
    * Levodopa; or
    * Drugs which alter GI pH/movement (e.g., omeprazole, ranitidine).
34. Use of vaccine including COVID-19 vaccine within 14 days prior to the first drug administration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Uncorrected and baseline-corrected sapropterin AUCt | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  The area under the analyte concentration versus time curve from time zero to the time of the last measurable analyte concentration (t)
Uncorrected and baseline-corrected sapropterin AUCinf | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  The area under the analyte concentration versus time curve from time zero to infinity
Uncorrected and baseline-corrected sapropterin Cmax | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  Maximum measured plasma analyte concentration over the sampling period

SECONDARY OUTCOMES:
Uncorrected and baseline-corrected sapropterin Tmax | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  Time of the maximum measured analyte concentration over the sampling period
Uncorrected and baseline-corrected sapropterin Tlag | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  Time of observation prior to the first observation with a measurable (non-zero) concentration

OTHER OUTCOMES:
Uncorrected and baseline-corrected sapropterin Thalf | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  The apparent elimination half-life
Uncorrected and baseline-corrected sapropterin Residual area | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  Percentage of AUC0-inf due to extrapolation from the time of the last observed concentration to infinity, calculated as [1 - (AUC0-t/AUC0-inf)] x 100
Uncorrected and baseline-corrected sapropterin Kel | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  Apparent first-order elimination rate constant
Uncorrected and baseline-corrected sapropterin Vz/F | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  Apparent Volume of Distribution
Uncorrected and baseline-corrected sapropterin CI/F | Pre-dose (-1, -0.5, and 0-hour) and at 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours post-dose (22 time points)
  Apparent clearance
Evaluate the Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Safety monitored from the signature of the Informed Consent through study completion (approximately 10 days)
  AEs will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA).

CONTACTS AND LOCATIONS:
Overall Officials: Mark L. Freedman, MD,FRCPC, Principal Investigator — Canada, Ontario - Pharma Medica Research Inc. 4770 Sheppard Ave E